CLINICAL TRIAL: NCT06495320
Title: Effect of Rational Drug Education on the Attitudes of Parents of Hospitalized Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Aslı Akdeniz Kudubeş, ASSOCIATE PROFESSOR, Bilecik Seyh Edebali Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: BILECIKSEYHEDEBALIUNIVERSITY
Record Dates: First submitted 2024-07-01; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Nursing Caries
Keywords: Rational drug use; Hospitalized Children; Parents
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: A parallel group (experiment-control) randomized controlled design, which is one of the experimental methods
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Rational drug use education will be applied to the experimental group.
  Interventions: Other: Rational drug use education
- Control group (No Intervention): No action will be taken

INTERVENTIONS:
Other: Rational drug use education — Rational Drug Use Education Program for Parents: The training program consists of 30 minutes. The training program will be delivered to parents in the form of a 30-minute training session with a powerpoint presentation, using the face-to-face education model. Interactive education methods that enable parents' participation will be used. In addition, in order to increase the permanence of education, the educational content will be given to parents in the form of an educational booklet.
  Other Names: education
  Arms: Experimental group

SUMMARY:
In this project, it was aimed to determine the effect of the rational drug management training program on parents' attitudes towards rational drug use. The project is designed as a randomized controlled study and will consist of experimental and control groups. An education program on rational drug use will be applied to the parents in the experimental group. The originality of this project is the evaluation of the effect of the education program on rational drug use applied to parents whose children are hospitalized. Although studies on rational drug use in parents have increased in recent years, most of them consist of descriptive studies aimed at evaluating knowledge and attitudes towards rational drug use. It seems that the number of intervention studies on rational drug use in parents is limited. No intervention studies aimed at the rational drug use attitudes of parents whose children are hospitalized have been found. This study has the feature of revealing the effectiveness of the rational drug use education program to be applied to parents in cases of illness and hospitalization where the importance of rational drug use becomes evident.

DETAILED DESCRIPTION:
The aim of the research will be carried out using a parallel group (experiment-control) randomized controlled design, which is one of the experimental methods, to determine the effect of the rational drug management training program on parents' attitudes towards rational drug use.

Goals:

* To examine the effect of the rational drug management training program on parents' attitudes towards rational drug use,
* To compare the average scores of the attitude scale towards rational drug use between the parents in the experimental group and the control group in the project.

ELIGIBILITY:
Inclusion Criteria:

* Having a child between the ages of 0-12,
* admitted to the pediatric ward,
* who have not previously received training on rational drug use
* Parents who volunteered to participate in the study

Exclusion Criteria:

* illiterate
* parents with mental retardation, vision and hearing impairment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Parental Attitude Scale Towards Rational Drug Use mean score | up to 10 months
  The effect of the applied education on the mean score of the Parental Attitude Scale Towards Rational Drug Use will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: BİLECİK ŞEYH EDEBALİ UNIVERSITY, Study Director — BİLECİK ŞEYH EDEBALİ UNIVERSITY
Locations (1):
- Asli Kudubeş, Bilecik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No